CLINICAL TRIAL: NCT00942617
Title: Measurement of Platelet Dense Granule Release in Healthy Volunteers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding issue
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Oates, Professor of Medicine and Pharmacology, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB# 080895; NIH/NHLBI #81009
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Platelet Aggregation
Keywords: platelet aggregation; granule secretion; thromboxane production; cyclooxygenase-1; ATP release; aspirin resistance; platelet activation; flow cytometry; Platelet aggregation in healthy volunteers
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 40 mg non-enteric coated aspirin (Experimental): 40 mg non-enteric coated ASA once daily for 21 + or - 2 days
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 40 mg non-enteric coated ASA once daily for 21 + or - 2 days

SUMMARY:
Aspirin has been shown to reduce cardiovascular events in at risk individuals. Elucidation of mechanisms of aspirin resistance and a possible loss of effect of aspirin over time with chronic aspirin treatment necessitate a more precise method of measuring the "release phase" of platelet activation, including the release of dense granules from platelets.

DETAILED DESCRIPTION:
This is a proposal for a pilot study to evaluate the feasibility of measuring 5-hydroxytryptamine (5-HT) release from platelets as an indicator of dense granule release during platelet activation in volunteers taking aspirin.

One phase of platelet response to activating agonists involves release of dense granules, which are known to contain 5HT (serotonin) and ATP. There are various methods of measuring the degranulation of platelets: ATP release can be measured using a lumiaggregometer, and release of 14C radiolabeled 5-HT from platelets. Using the aggregometer and a 14C labeled 5-HT assay can be used to measure 5-HT release from platelets.

Our experience suggests that ADP-induced ATP release is insensitive to detect very low levels of platelet dense granule release, which occurs in aspirin-treated subjects. The pilot study will permit optimizing the method for reliably detecting low levels of 5HT release in patients who achieve submaximal inhibition of the cyclooxygenase during aspirin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males over age 18
* Non-smokers
* No chronic medical illness
* No chronic medications

Exclusion Criteria:

* ASA/NSAID use previous 14 days.
* History of chronic NSAID use.
* Currently taking NSAIDs, opioid analgesics, corticosteroids, or anticoagulants.
* History of coronary artery disease, myocardial infarction, coronary artery bypass grafting, percutaneous angioplasty, diabetes mellitus or stroke.
* History of hypertension
* BMI >35
* Smokers
* History of gastric, duodenal, or esophageal ulcers or serious gastrointestinal bleed.
* History of frequent headaches, pain syndrome, or other condition requiring frequent use of analgesics.
* History of adverse reaction to ASA.
* Initial platelet count <100K/µl or >500K/µl.
* Initial hematocrit <35% or >50%.
* Weight less than 110 pounds.

Female subjects will be excluded to avoid possible confounding uterine smooth muscle production of prostaglandins which various throughout the menstrual cycle.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary measurement will be platelet 5-HT release induced by ADP after 1 and 2 weeks administration of daily ASA. | 3 weeks

SECONDARY OUTCOMES:
Measurements will include platelet COX-1 activity, flow cytometric measurement of markers of platelet activation, platelet aggregation and ATP release, and serum thromboxane B2 (TxB2) levels, at each timepoint. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John A Oates, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States